CLINICAL TRIAL: NCT05409014
Title: Effect of Pelvic Floor Muscle Training on Urinary Incontinence Symptoms and Quality of Life in Women Who Practice Physical Exercise
Brief Title: Pelvic Floor Muscle Training on Urinary Incontinence Symptoms and Quality of Life in Women Who Practice Physical Exercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of the State of Santa Catarina (Other)
Responsible Party: Principal Investigator, Gilmar Moraes Santos, PT, Clinical Professor, University of the State of Santa Catarina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PFMT exercise
Record Dates: First submitted 2022-06-02; First posted 2022-06-07 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Urinary Incontinence; Pelvic Floor Disorders; Quality of Life
Keywords: Pelvic Floor; Exercise
MeSH Terms: conditions — Urinary Incontinence; Pelvic Floor Disorders; Motor Activity

STUDY DESIGN:
Intervention Model Description: This was a single-group clinical trial evaluating the effect of pelvic floor muscle training in incontinent women who exercise.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PFMT (Experimental): The exercises of this protocol were performed at home, but with face-to-face meetings in the first phase of the protocol (awareness) and every 15 days, where the physical therapist taught the new exercises to be performed in the next phase. All protocol meetings were performed by a trained physical therapist/researcher. In situations where it was not possible to hold the meetings in person, due to the Covid-19 pandemic, they were held online through video calls with the responsible researcher. The PFMT protocol lasts for eight weeks and was divided into five phases: awareness, stabilization, strength, potency and potency complement. Each phase is 2 weeks long.
  Interventions: Other: PFMT

INTERVENTIONS:
Other: PFMT — The phase 1 of the protocol was awareness-raising, the athlete receives guidance from a physical therapist and learns the location of the PFM and the ability to contract them in isolation. The phase 2 is stabilization, consisting of 15 stabilization exercises, which are performed through pelvic floor contractions for 10 seconds and with the same relaxation time, repeating each group 10 times. The phase 3 is strength, the same exercises as the second phase are performed using 2 kg weights at the end of each leg and/or arm. There are eight groups of exercises and with changes in the time of slow contraction and relaxation. The phase 4 is power, in power exercises the training loads are increased and the sequence of movements is also increased. The phase 5 is to complement the power, this phase was the continuation of the previous one in the sense of potentiation of the results where ballistic movements, speed and impact fundamentally predominate.

SUMMARY:
Introduction: The practice of physical exercises can lead to the development of urinary incontinence (UI) symptoms, in addition to negatively impacting the function of the pelvic floor muscles (PFM) and the quality of life (QoL) of women. Aim: To evaluate the effect of pelvic floor muscle training (PFMT) on UI symptoms and QoL in women who practice physical exercise. Methods: The clinical trial was carried out in two stages, one online and the other in person. The online stage was carried out through a website, with the application of forms and validated questionnaires on urine leakage (International Consultation on Incontinence Questionnaire - Short Form) and quality of life (King's Health Questionnaire). In the face-to-face interview, all women practicing physical exercise and with symptoms of UI were invited to perform PFM assessment and Pelvic Organ Prolapse - Quantification (POP-Q) System, then the PFMT protocol. Women aged 18 years or older, in the reproductive phase and who practiced regular physical exercise for at least 6 months and at least 3 times a week were included. Results: Women are expected to improve UI symptoms and quality of life after PFMT.

DETAILED DESCRIPTION:
This is a non-randomized controlled clinical trial. The present research was approved by the Ethics Committee in Research with Human Beings of the Universidade do Estado de Santa Catarina (UDESC) with number 4.670.454. Data collection took place between November 2021 and June 2022 in two stages, one online and the other in person. The online stage was carried out through a website developed by the research team (https://projetocrossfititudesc.wixsite.com/saudedamulher), on this website the participants agreed to the Free and Informed Consent Term; completed forms on sociodemographic data, presence of UI and urinary habits and their participation in physical exercise; and completed validated questionnaires on urine leakage (International Consultation on Incontinence Questionnaire - Short Form) and quality of life (King's Health Questionnaire).

In the face-to-face stage, all women who practiced physical exercise and had symptoms of UI were invited to undergo an evaluation of the PFM and, then, the PFMT protocol at the Biomechanics Laboratory of the Center for Health Sciences and Sport (CEFID/UDESC). This protocol lasted eight weeks and consisted of five phases. At the end of the eight weeks, the same forms, questionnaires and PFM evaluation procedures were applied by the same evaluator.

All participants were recruited through the dissemination of a folder on social media (Instagram, Whatsapp and through the UDESC website) and visits to the exercise practice places (gyms and Crossfit box).

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years of age;
* Practitioners of any physical exercise for at least six months and with a frequency of at least three times a week.

Exclusion Criteria:

* Women with climacteric or menopausal symptoms;
* Who report symptoms of urinary tract infection in the last week (self-reported pain and burning sensation when urinating);
* Who underwent physiotherapeutic, surgical or drug treatment in the last 6 months for UI;
* Diagnosis or signs and symptoms of ongoing neurological, cardiac, gastrointestinal or genitourinary diseases;
* Being in the gestational period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-05-13 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Urinary incontinence symptoms | Pre intervention and 8 week post intervention
  Will be assessed using the International Consultation on Incontinence Questionnaire - Short Form (ICIQ-UI SF). It is a simple, brief (four-item) and self-administered questionnaire that asks the frequency of urine leakage (0 = "Never" to 5 = "All the time"), the volume of urine lost (0 = "None" to 6 = "A large amount") and the impact of UI on quality of life (0 = "Does not interfere" to 10 = "It interferes a lot"). For women undergoing non-surgical treatments for UI, 4-point reductions in the overall ICIQ-UI SF score are perceived as clinically significant (LIM et al., 2019). The fourth item has eight alternatives with situations in which the individual may have urine leakage and aims to identify the type of UI.

SECONDARY OUTCOMES:
Quality of life | Pre intervention and 8 week post intervention
  The King's Health Questionnaire assesses the impact of UI on different domains of quality of life and perceived symptoms. It consists of 21 questions divided into 8 domains (general health perception, impact of UI, limitations of daily activities, physical limitations, social limitations, personal relationships, emotions and sleep/disposition) and two independent scales (measures of severity and scale of urinary symptoms). The score is calculated as a percentage per domain.The higher the percentage, the greater the impact of UI on quality of life.
Maximal voluntary contraction | Pre intervention and 8 week post intervention
  Peritron 9300® manometer will be used to assess the maximum voluntary contraction (MVC). An MVC of PFM will be asked to the participant and the peak value was recorded, this process was repeated 3 times. The mean value of these three pressure peaks corresponded to MVC of the PFM.
Vaginal resting pressure | Pre intervention and 8 week post intervention
  Peritron 9300® manometer will be used to assess the vaginal resting pressure (VRP). For the assessment of VRP, a command was given to the participant to relax the PFM and then given a rest period to control the influence of possible voluntary and involuntary contractions, in order to obtain the measure of VRP.
Pelvic Organ Prolapse - Quantification (POP-Q) System | Pre intervention and 8 week post intervention
  The Pelvic Organ Prolapse - Quantification (POP-Q) System is a system used to describe, quantify and maintain pelvic support in women. Specific points that are considered when recording the POP-Q and as measurements expressed in centimeters. Positive values refer to positions below or distal to the hymen (reference point), negative values above or proximal to the hymen, and the hymen plane is set to zero. The six points are located on the anterior, superior and posterior wall of the vaginal canal. Other measurements include the genital hiatus, the perineal body, and the total length of the vagina. All points are average at most, except total vaginal compliance. The application provided by the American Urogynecologic Society was used to score the measurements and correctly classify the POP grade into: grade 0, grade I, grade II, grade III or grade IV.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Ciências da Saúde e do Esporte (CEFID), Florianópolis, Santa Catarina, Brazil